CLINICAL TRIAL: NCT07379346
Title: Investigation of the Effect of Virtual Reality Assisted Exercise Program on Physical Parameters in Hockey Players: Single Blinded Randomize Controlled Trial
Brief Title: Investigation of the Effect of Virtual Reality Assisted Exercise Program on Physical Parameters in Hockey Players
Acronym: VRHOCKEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Ertugrul Deniz Kose, Assist. Prof. Dr., Amasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amasya Uni-E.10568
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Virtual Reality Based Therapy; Ankle Dorsiflexion; Motor Learning; Agility
Keywords: Assistive Technology; Balance Control; Motor Learning; Sensorimotor Integration; Virtual Reality

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups. The control group continues routine hockey training only, while the intervention group continues routine training and additionally receives a virtual reality-assisted exercise program. Group allocation remains fixed throughout the study, and outcomes are compared between groups across three assessment time points (baseline, post-intervention, and follow-up).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments are performed by a physiotherapist who is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Hockey Training (Control) (No Intervention): Participants continue routine hockey training (warm-up, passing drills, offense-defense organization, penalty-corner practices) 3 days/week.
- Routine Training + VR-Assisted Exercise (Experimental): Participants continue routine hockey training and additionally perform virtual reality-assisted exercises using the Nintendo Wii Balance Board, 30 minutes/session, 3 sessions/week, for 6 weeks.
  Interventions: Device: Nintendo Wii Balance Board Exergaming

INTERVENTIONS:
Device: Nintendo Wii Balance Board Exergaming — Obstacle Course, Ski Slalom, and NFL Slapshot; 30 minutes/session; 3 sessions/week; 6 weeks.
  Arms: Routine Training + VR-Assisted Exercise

SUMMARY:
This single-blind randomized controlled trial investigates the effects of a virtual reality-assisted exercise program added to routine hockey training on balance, functional ankle dorsiflexion, agility, and shooting performance in youth hockey players. Participants are randomly assigned to either routine training alone or routine training plus a 6-week virtual reality-assisted exercise intervention delivered via the Nintendo Wii Balance Board. Outcomes are assessed at baseline, post-intervention, and at 3-week follow-up by a blinded assessor.

DETAILED DESCRIPTION:
This study is designed as a single-blind randomized controlled trial to evaluate the effects of a virtual reality-assisted exercise program on balance, functional ankle dorsiflexion, agility, and shooting performance in youth hockey players. Participants are recruited from a competitive hockey team and randomly assigned to either a control group or an intervention group.

The control group continues routine hockey training, including warm-up exercises, passing drills, offense-defense organization, and penalty-corner practices, three days per week. The intervention group continues the same routine training and additionally participates in a virtual reality-assisted exercise program delivered via the Nintendo Wii Balance Board. The virtual reality intervention includes Obstacle Course, Ski Slalom, and NFL Slapshot games and is administered for 30 minutes per session, three sessions per week, over a 6-week period.

Outcome measures include dynamic balance assessed by the Y Balance Test, agility assessed by the T-run agility test, functional ankle dorsiflexion assessed by the weight-bearing lunge test, and shooting performance assessed using a standardized target-based shooting accuracy protocol. All outcomes are assessed at baseline, immediately after the 6-week intervention period, and at a 3-week follow-up. Outcome assessments are performed by a physiotherapist who is blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Youth hockey players affiliated with a competitive hockey team
* Aged between 16 and 25 years
* Regular participation in routine hockey training
* Voluntary participation with written informed consent

Exclusion Criteria:

* Presence of an injury preventing participation in routine hockey training
* Presence of visual or neurological conditions that may interfere with virtual reality-assisted exercises
* Failure to attend the virtual reality-assisted exercise program for more than two consecutive sessions

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Shooting Performance | Baseline, immediately post-intervention (6 weeks), and 3-week follow-up
  Shooting performance is assessed using a standardized target-based shooting accuracy protocol. Participants perform drag-flick shots toward predefined target zones, and total hit scores are recorded. Higher scores indicate better shooting accuracy.

SECONDARY OUTCOMES:
Dynamic Balance (Y Balance Test) | Baseline, post-intervention (6 weeks), and 3-week follow-up
  Dynamic balance is evaluated using the Y Balance Test. Normalized reach distances are recorded for each limb.
Functional Ankle Dorsiflexion (Weight-Bearing Lunge Test) | Baseline, post-intervention (6 weeks), and 3-week follow-up
  Functional ankle dorsiflexion is assessed using the weight-bearing lunge test, with dorsiflexion angle measured for both ankles.
Agility (T-run Agility Test) | Baseline, post-intervention (6 weeks), and 3-week follow-up
  Agility is assessed using the T-run agility test, with performance recorded as completion time in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul Deniz KÖSE, Ph.D, Principal Investigator — Amasya University
Locations (1):
- Amasya University, Amasya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in this study will be available from the corresponding author upon reasonable request, following publication. Requests will be reviewed to ensure appropriate use and compliance with ethical approvals.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From publication
Access Criteria: Access to the de-identified individual participant data will be granted to qualified researchers upon reasonable request, subject to approval by the corresponding author and in compliance with ethical approvals.

REFERENCES:
- [Background] Polikanova I, et al. Virtual reality training improves balance and agility in athletes. Journal of Sports Sciences. 2021;39(4):456-464. Laufer Y, et al. The effect of virtual reality-based training on postural control. Gait & Posture. 2014;40(2):285-291. Schmitt KU, et al. Balance and sensorimotor training in sports performance. Sports Medicine. 2019;49(3):421-435.